CLINICAL TRIAL: NCT02014766
Title: A Randomized Comparison of Ultrasound-guided Supraclavicular and Interscalene Block After Shoulder Surgery
Brief Title: Supraclavicular Versus Interscalene Block
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cheju Halla General Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Inter1; 2013-M10 (Other: Cheju Halla General Hospital)
Record Dates: First submitted 2013-12-06; First posted 2013-12-18 (Estimated); Last update posted 2013-12-18 (Estimated); Status verified 2013-12

CONDITIONS: Pain
MeSH Terms: conditions — Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Interscalene block (Active Comparator): Interscalene block is performed under ultrasound guidance. Linear probe is placed on the ipsilateral interscalene groove visualizing the brachial plexus located between anterior and middle scalene muscles. Using in-plane technique, an insulated needle is advanced into the brachial plexus sheath, into which 20 ml of 0.375% ropivacaine is injected.
  Interventions: Procedure: Interscalene block
- Supraclavicular block (Experimental): Supraclavicular block is performed under ultrasound guidance. Linear probe is placed on the ipsilateral supraclavicular fossa visualizing the brachial plexus located lateral to the subclavian artery. Using in-plane technique, an insulated needle is advanced into the brachial plexus sheath, into which 20 ml of 0.375% ropivacaine is injected.
  Interventions: Procedure: Supraclavicular block

INTERVENTIONS:
Procedure: Interscalene block — Ultrasound-guided interscalene block is performed.
  Arms: Interscalene block
Procedure: Supraclavicular block — Ultrasound-guided supraclavicular block is performed
  Arms: Supraclavicular block

SUMMARY:
We hypothesize that both ultrasound-guided supraclavicular and interscalene block provide similar analgesia after shoulder surgery.

DETAILED DESCRIPTION:
Interscalene block provides effective postoperative analgesia after shoulder surgery. However, it can be associated with significant risk including the phrenic nerve palsy. Previous study reported that ultrasound-guided interscalene and supraclavicular blocks are effective and safe for shoulder arthroscopy.

ELIGIBILITY:
Inclusion Criteria:

American Society of Anesthesiologists physical status I-III inpatients undergoing shoulder surgery

Exclusion Criteria:

pregnancy, severe respiratory disease, preexisting neuropathy in the operated arm, coagulopathy, allergy to study medication

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2013-11; Primary Completion 2014-12 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
pain duration | at 24h after operation

SECONDARY OUTCOMES:
diaphragmatic movement | preoperative, after block(at 30 min), after operation
motor block | after block(at 30 min), after operation, at 24h
paresthesia | after block(at 30min), after operation, at 24h
complications | after block (at 30 min), after operation, at 24h
supplemental analgesia | after operation, at 24h
pain score | at 24h
patient satisfaction | at 24h

CONTACTS AND LOCATIONS:
Overall Officials: Chunwoo Yang, MD, Principal Investigator — Dep. of anesthesia and pain medicine, Cheju Halla General Hospital
Locations (1):
- Cheju Halla General Hopsital, Jeju City, Jeju Self-governing Province, South Korea

REFERENCES:
- [Background] Fredrickson MJ, Krishnan S, Chen CY. Postoperative analgesia for shoulder surgery: a critical appraisal and review of current techniques. Anaesthesia. 2010 Jun;65(6):608-624. doi: 10.1111/j.1365-2044.2009.06231.x. PMID 20565394
- [Result] Liu SS, Gordon MA, Shaw PM, Wilfred S, Shetty T, Yadeau JT. A prospective clinical registry of ultrasound-guided regional anesthesia for ambulatory shoulder surgery. Anesth Analg. 2010 Sep;111(3):617-23. doi: 10.1213/ANE.0b013e3181ea5f5d. Epub 2010 Aug 4. PMID 20686013